CLINICAL TRIAL: NCT06656819
Title: TMSpine: The Modulatory Effect of Female Sex Hormones on Spinal Neuroplasticity
Brief Title: The Modulatory Effect of Female Sex Hormones on Spinal Neuroplasticity
Acronym: TMSpine
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Yasin Dhaher, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2020-0738
Record Dates: First submitted 2024-08-21; First posted 2024-10-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Healthy Females
  Interventions: Device: Magstim Rapid2
- Healthy Males (control)
  Interventions: Device: Magstim Rapid2

INTERVENTIONS:
Device: Magstim Rapid2 — AIM 1: Investigate the estradiol effect on spinal circuit excitability post afferent (sensory) mediated subthreshold motor priming in young healthy women and men.
  AIM 2: Characterize the Input output property of spinal circuit excitability following descending drive (motor) mediate priming in young healthy participants
  AIM 3: Examine the estradiol effect on spinal circuit excitability following descending drive (motor) mediated priming in young healthy females

SUMMARY:
The goal of this project is to test our central hypothesis that the spinal cord neuroplasticity in females will be modulated by the level of estradiol concentration. under aim 1 we will determine the influence of estradiol fluctuations on spinal circuit excitability post afferent (sensory) mediated subthreshold motor priming in young healthy females and males. We will use an established repetitive peripheral nerve electrical stimulation with a stimulation intensity below the motor threshold to prime the spinal motor circuits. under aim 2 we seek to characterize the input output property of spinal circuit excitability after descending drive (motor) mediated priming in young healthy male participants. in aim 3 we will examine the influence of estradiol fluctuations on descending drive mediated motor priming in young healthy females.

ELIGIBILITY:
FEMALES

Inclusion Criteria:

* Ages 18-39 years
* Eumenorrheic (regular monthly cycles of 24-35 days)
* Moderately active (less than 7 hours of vigorous physical activity per week)
* History of pregnancy is allowed if patient is in post-lactation phase

Exclusion Criteria:

* History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot
* History of neurological injury of the peripheral or central nervous system
* Current smoker
* History of disordered eating
* History of stress fracture in the lower limb
* History of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease)
* Pacemaker, metal implants in the head and spine region
* Pregnancy
* On a hormonal contraceptive regimen (oral, transdermal or vaginal)
* History of menstrual dysfunction (primary or secondary amenorrhea, oligomenorrhea, anovulatory cycles, polycystic ovarian disease)
* Started or stopped taking oral contraceptives within the previous 6 months
* Exercise vigorously more than 7 hours per week or currently participating in competitive level sports.

MALES

Inclusion Criteria:

* Ages 18-39
* Moderately active (less than 7 hours of vigorous physical activity per week)

Exclusion Criteria:

* History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot
* History of neurological injury of the peripheral or central nervous system
* Current smoker
* History of disordered eating
* History of stress fracture in the lower limb
* History of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease)
* Pacemaker, metal implants in the head and spine region

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: (1) Healthy females (2) Healthy males (control)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Spinal circuit excitability | Baseline 1, Post-60mins after peripheral nerve stimulation
  Change in Spinal circuit excitability will be assessed by measuring Hoffmann reflex/ M wave ratio of the soleus muscle. Higher scores indicate poorer outcome.
Change in Motor neuron excitability | Baseline 2, Post-60mins after priming
  Changes in motor neuron excitability, as quantified by Delta-F values.
Change in spinal reflex expression | Baseline 2, Post-60mins after priming
Change in descending drive mediated motor priming | Baseline 2, Post-60mins after priming

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Dhaher, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States